CLINICAL TRIAL: NCT05400161
Title: Social Media-Based Parenting Program for Women With Postpartum Depressive Symptoms
Brief Title: Social Media-Based Parenting Program for Women With Postpartum Depressive Symptoms: Impact on Child Development
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-019784; R33MH118405 (NIH)
Record Dates: First submitted 2022-05-27; First posted 2022-06-01 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Postpartum Depression; Parenting; Parent-Child Relations; Child Development
Keywords: Social Media; Parenting; Postpartum Depression; Mothers; Infants; Childhood Developmental Outcomes; Postpartum; Depression; Mother-Infant Interactions
MeSH Terms: conditions — Depression, Postpartum; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Video coders will be blinded to intervention assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MoodGym Alone (Active Comparator): The MoodGym program is an evidence-based online cognitive behavioral treatment program that has been shown to be effective at reducing depression symptoms in a meta-analysis of 11 trials (g=0.36, 95% CI 0.17-0.56). Moodgym contains five modules with interactive exercises, workbooks, anxiety and depression quizzes, and downloadable relaxation audio files that can be completed online without therapist interaction.
  Interventions: Behavioral: MoodGym
- Parenting Program + MoodGym (Experimental): The social media-based parenting program consists of 8 weekly sessions using a Facebook platform with the following topics: depression psychoeducation and behavioral activation, infant temperament, play, feeding, safety, sleep, parent-child interactions, and shared book reading. Participants in the experimental arm will also be enrolled in the online depression treatment program, MoodGym.
  Interventions: Behavioral: MoodGym; Behavioral: Social Media-Based Parenting Program

INTERVENTIONS:
Behavioral: MoodGym — Participants in the control group will be enrolled in MoodGym, an evidence-based online Cognitive Behavioral Therapy (CBT) program for depression. Through the MoodGym program, participants will have access to interactive exercises, workbooks, anxiety and depression quizzes, and downloadable relaxation audio files. Investigators will supplement Moodgym with a facilitator contact by texting or email to check-in and encourage completion of intervention. MoodGym will provide information on the number of sessions completed by participants (engagement and dosage).
Behavioral: Social Media-Based Parenting Program — Participants in the intervention group will be enrolled in Facebook secret user groups, administered by a trained facilitator, to permit participants to view and comment on posted materials. Content and user identity are restricted to invited participants to maintain privacy. Investigators will organize educational materials into video vignettes, narrated PowerPoint presentations, and written materials. The facilitator reviews and comments on postings daily and provides feedback to participants. Facebook analytics for the secret groups are available to group administrators and will provide information on any sessions viewed and counts of sessions viewed and comments posted. Participants randomized to the intervention will also have the option to take part in a preliminary virtual session through a secure video platform (e.g. BlueJeans) and will receive weekly engagement text messages. Women in the intervention group will be enrolled in the online depression treatment program, MoodGym.
  Arms: Parenting Program + MoodGym

SUMMARY:
The long-term goal is to develop effective parenting strategies to facilitate optimal child development for mothers suffering with PPD symptoms. The overall objective for this application is to study whether this program combined with online depression treatment leads to more responsive parenting (target) and signals improved child language, socioemotional and cognitive development (outcomes) compared to depression treatment alone. Findings from this application can be used to inform a future study to test the effectiveness and implementation of this social media-based parenting program.

DETAILED DESCRIPTION:
Postpartum depression (PPD) symptoms are common among women following the birth of a child and can adversely impact a mother's ability to care for her child. As a result, infants of mothers with PPD symptoms may experience less responsive parenting, placing them at greater risk for delays in development. Evidence- based parenting programs have been developed to guide mothers with caring for their infants but may not address the impact of depression on parenting, are intensive and expensive to administer with limited ability for scale up, or are not available in a format that facilitates participation by women with depressive symptoms. To address these barriers, investigators developed a theoretically-driven social media-based parenting program on responsive parenting and child development.

To determine whether the social media-based parenting program can improve responsive parenting and signal greater child development among women with PPD symptoms, investigators will conduct a prospective individually randomized group treatment trial. 113 eligible women who screen positive for PPD at their infants' well child visit and their children will be consented, enrolled, and randomized as mother-child dyads 1:1 to receive a) the social media-based parenting program plus online depression treatment or b) online depression treatment alone. Investigators chose a randomized design, because it is most effective in guarding against bias and will ensure that patients in both arms are similar in observed and unobserved characteristics. Treatment assignment will be done at the time of enrollment following informed consent.

Descriptive statistics for demographic and poverty characteristics and PPD symptoms measured at baseline will be examined across the two treatment groups to assess the success of the randomization. Investigators will assess responsive parenting at baseline and 3 months post-enrollment. Secondary endpoints which include the changes in EPDS, PSOC, and PSI-SF scores measured between baseline and the 3-month follow-up between groups, will be explored to determine if the effects of the parenting program are consistent with preliminary study findings. The secondary child developmental outcomes will include differences in the Bayley-3 cognitive, language, and motor subscale scores at the 12-month follow-up visit. The intervention arm will also be assessed with the Therapeutic Factors Inventory-8 (TFI-8) to measure cohesion and the Acceptability survey which measures feasibility of the parenting program at 3-months post-enrollment. Additionally, at the 3-month mark, all participants will be administered the MoodGym Acceptability Survey to assess feasibility of the online depression treatment program.

The results of this application would be expected to contribute important new knowledge and inform a future trial on parenting strategies to better assist mothers with PPD symptoms and improve child developmental outcomes.

ELIGIBILITY:
Inclusion Criteria:

Women who:

* Are >18 years old
* Screen positive for postpartum depression (score>9) on the EPDS at a -participating pediatric practice
* Have an infant <8 months of age
* Speak and Read English
* Have Access to a smart phone or computer tablet with internet access

Children who:

-Are < 8 months old

Exclusion Criteria:

Women who:

* Report suicidality (i.e., suicidal ideation and/or behavior) on the EPDS (Question #10) at enrollment.
* Report severe depressive symptoms (EPDS>20) at enrollment.
* Have a substantiated report of child maltreatment

Children who:

* Were born premature (estimated gestational age<35 weeks)
* Have been diagnosed with congenital malformations or genetic syndromes which place them at risk of developmental delays
* Are already currently receiving early intervention services for developmental delays at baseline

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2022-11-18 (Actual); Primary Completion 2025-04-14 (Actual); Study Completion 2025-04-14 (Actual)

PRIMARY OUTCOMES:
Changes in parent-child interactions | Baseline and 3-months
  The Parent Child Early Relational Assessment (PCERA) will be used to assess parent-child interactions. The PCERA is a validated 65-item videotape assessment designed to measure the quality of affect and behavior in parent-infant interactions. The PCERA uses ratings that are based on observations of 5-minute videotaped interactions with parent-infant dyads engaged in free play. The PCERA contains 8 subscales of which 3 parenting subscales will be the focus: 1) Parental Positive Affective Involvement and Verbalization, 2) Parental Negative Affect and Behavior, and 3) Parental Intrusiveness, Insensitivity, and Inconsistency. Each individual subscale is scored between 0-5, with higher scores indicating more responsive parenting. A subscale score of 1-2 indicates an area of concern, a score of 3 indicates some concern, and a score of 4-5 in

SECONDARY OUTCOMES:
Changes in severity of depressive symptoms | Monthly (Baseline to 12-months)
  Severity of depressive symptoms will be measured by using the Edinburgh Postnatal Depression Scale (EPDS). The EPDS is a validated 10-item self-report measure of depressive symptoms with strong evidence for reliability, validity, and utility in varying populations. It has been used extensively in mental health research and provides cutpoints to determine the severity of depressive symptoms. It includes a question on suicidal thoughts and wishes (#10) that will be used to monitor for suicidality. The total score (range: 0-30) will be used with scores of 10 or higher representing minor or moderate depression and scores of 20 or greater representing severe depression.These outcomes will assess changes in EPDS from baseline to 3 months.
Changes in parenting competence | Baseline and 3-months
  Parenting competence will be measured using the Parenting Sense of Competence Scale (PSOC). The PSOC is a validated 17-item self-report measure of parenting self-esteem and competence and consists of two factors: satisfaction and efficacy. Response categories are on a 6-point likert-scale from strongly disagree to strongly agree. The total score (range: 17-102), which includes the sum of the two factors, will be used. A higher score indicates a higher parenting sense of competency. There are no average scores or 'cut-off's' for this tool. These outcomes will assess changes in PSOC from baseline to 3 months.
Changes in parenting stress | Baseline and 3-months
  Parenting stress will be measured using the Parenting Stress Index-Short Form (PSI-SF). The PSI-SF is a validated 36-item scale that measures parenting stress. The PSI-SF is a direct derivative of the full-length test (PSI) and it has been shown to have excellent internal consistency and to be positively associated with maternal psychological distress. Scores on the PSI-SF correlate well with the full-length PSI. It yields a Total Stress score from three scales: Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child. The total score (range: 36-180) will be used, with higher scores indicating higher levels of stress.These outcomes will assess changes in PSI-SF from baseline to 3 months.
Prior mental health service use | Monthly (Baseline to 12-months)
  Prior mental health service use will be measured using the National Comorbidity Survey (NCS), which provides data on mental health treatment in the United States. Investigators will include a question from the NCS on prior mental health services use in the past month: "In the past month, did you receive treatment for problems with your emotions or nerves, or your use of alcohol or drugs?" We will consider mental health service use to have occurred in the past month if a mother responds "Yes" to this question. The results indicate the number of participants from each group who received mental health services/treatment at each time point. Additionally, if a mother responds "Yes" to the initial NCS item, a follow-up question will be asked to determine the specific types of services that were accessed: "If yes, what type of treatment did you receive?"
Social support | Baseline
  Social support will be measured using the Multi-dimensional Scale of Perceived Social Support (MSPSS). The MSPSS is a 12-item scale that assesses perceived social support from family, friends, and a significant other. Response categories are on a 7-point likert-scale from 1=very strongly disagree to 7=very strongly agree. The total score will be used (range: 12-84).
Therapy group cohesion | 3-months
  Therapy group cohesion will be measured using the TFI-8. The TFI-8 is a validated 8-item scale that is used to measure cohesion and is continuous process monitoring for therapy groups. Scores on the TFI-8 correlate well with the full TFI. The total score (range: 8-56) will be used, with higher scores indicating greater cohesion within the group. The TFI-8 will be administered at the 3-month visit to the intervention group, only.
Acceptability of the parenting program | 3-months
  Acceptability of the parenting program will be measured using the Acceptability Survey. The Acceptability Survey is a 10-item scale with 3 additional open ended questions. The total score (range: 9-45) will be used and the open ended questions will be qualitatively analyzed to help inform the acceptability scores. Higher scores on the acceptability survey indicate greater satisfaction and feasibility of the parenting program. The acceptability survey will be administered at the 3-month visit to the intervention, only.
Acceptability of the online depression treatment program | 3-months
  The acceptability of the online depression treatment program, MoodGym, will be measured using the MoodGym Acceptability Survey. The survey includes two qualitative open-ended questions and an additional question that asks, "It is ___________ that I will use MoodGym compared to going to a health care provider for depression treatment." The response is a 5-point likert-scale from "Much More Likely" to "Much Less Likely". The open ended questions will be qualitatively analyzed to help inform the acceptability scores. The MoodGym Acceptability survey will be administered at the 3-month visit to all participants.
Child Development | 12-months
  Child development will be measured using the Bayley Scales of Infant and Toddler Development-3rd Edition (BSID-III). The BSID-III is a validated scale of child development from 1 to 42 months of age. The BSID-III has excellent reliability and correlates well with other measures of development including the Wechsler Preschool and Primary Scale of Intelligence (r=0.83). The BSID-III has three subscales that will be utilized (cognitive, motor, and language).

CONTACTS AND LOCATIONS:
Overall Officials: James Guevara, MD,MPH, Principal Investigator — Children's Hospital of Philadelphia; Rhonda Boyd, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
A complete, cleaned, and de-identified dataset will be made available to other investigators after all analyses have been conducted and within twelve months of the end of the final year of funding to allow for publication of all study aims. To obtain this data set, other investigators will need to contact the study Principal Investigator (PI) who will provide a data sharing agreement. The data sharing agreement will permit a deidentified data set to be shared once an Institutional Review Board (IRB) protocol has been approved at the investigators' home institution and the investigators have signed a pledge to not attempt to identify individual study subjects. The data set will be made available on a Compact Disc Read-Only Memory (CD-ROM) or through a secure File Transfer Protocol (FTP) site.
Supporting Information: Study Protocol, SAP
Time Frame: 12 months after the end of the final year of funding.